CLINICAL TRIAL: NCT07334145
Title: Effect of SGLT2 Inhibitors On Anemia in Patients With Chronic Kidney Disease (CKD)
Brief Title: Effect of SGLT2 Inhibitors on Anemic CKD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Romany Nageb, resident of internal medicine at sohag university hospital, Sohag University
Other Study IDs: soh_med__25_12_6MS
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anemia in CKD Patients
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- CKD patients stage 1_4
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — prescription of SGLT2 inhibitors like dapagliflozin or empagliflozin to anemic CKD patients stage 1_4

SUMMARY:
anemia is a common complication of CKD patients and affect the quality of life and increase morbidity and mortality. managing anemia in CKD patients remains challenging conventional therapy including iron and ESAs which has its complications. the SGLT2 inhibitors have emerging evidence from major clinical trials in improving anemia in patients with CKD

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* CKD stage 1_4
* baseline hemoglobin 8.5 to 12.9 g/dl
* stable anemia regimen for more than 8 weeks

Exclusion Criteria:

* dialysis recent blood transfusion or ESA dose change within 8 weeks active malignancy or infection pregnancy or lactation history of recurrent DKA or sever volume depletion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people in sohag twen
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
hemoglobin level | 12 weeks
  use the hemoglobin level to assist the effect of SGLT2 inhibitors On anemia correction
change in hemoglobin level | 12 weeks
  anemia correction

CONTACTS AND LOCATIONS:
Overall Officials: Romany Naguib Mikhaeil, master, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Sohag University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided